CLINICAL TRIAL: NCT03068338
Title: Robotic Sock Technology for Prevention of Deep Vein Thrombosis and Joint Contracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: RSDVT001
Record Dates: First submitted 2017-02-26; First posted 2017-03-01 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-03

CONDITIONS: Deep Vein Thrombosis; Ankle Joint Contracture
MeSH Terms: conditions — Venous Thrombosis | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (Active Comparator): Intermittent pneumatic compression devices are used for prevention of DVT.
  Interventions: Device: Intermittent pneumatic compression
- Robotic Sock (Experimental): Soft robotic actuator used in a sock design technology to perform plantarflexion and dorsiflexion of the foot about the ankle joint.
  Interventions: Device: Robotic Sock

INTERVENTIONS:
Device: Robotic Sock — Soft robotic actuator used in a sock design technology to perform plantarflexion and dorsiflexion of the foot about the ankle joint.
  Arms: Robotic Sock
Device: Intermittent pneumatic compression — Conventional device used by hospitals
  Arms: Conventional therapy

SUMMARY:
The research team's aim is to investigate the effects of the team's soft robotic socks in providing assisted ankle dorsiflexion-plantarflexion and promoting venous blood flow in stroke patients. Specifically, the investigators intend to 1) observe the development of joint contracture in terms of the range of motion of the ankle joint given the use of the device 2) monitor the presence of blood clots in the deep veins using compression Duplex ultrasonography given the use of the sock device.

The investigators hypothesize that a soft robotics approach can provide compliant actuation to simulate natural ankle dorsiflexion and plantarflexion, which will consequently promote blood circulation in the lower leg of stroke patients who have not previously developed ankle joint contracture. This will prevent the occurrence of DVT and movement in the ankle joint will alleviate stiffness. This robotic sock intervention is to prevent the development of ankle joint contracture so established ankle contractures will be excluded from this study.

DETAILED DESCRIPTION:
The investigator's proposed robotic sock solution is capable of providing programmable robot-assisted ankle exercises to chronic bedridden patients, thereby improving venous blood flow, and preventing DVT and ankle joint contractures. Compared to conventional mechanical prophylaxis such as the intermittent pneumatic compression devices, the robotic sock is likely to cost almost five times less, and potentially generate patient/hospital savings of up to $2750 per patient. The use of the robotic sock will also raise therapist productivity through automating the therapy exercises of the bedridden patients, and this could potentially save the therapists at least 6 workhours per day. The use of the robotic sock in hospitals, nursing homes and patients' own homes will likely reduce healthcare costs and prevent side effects, as compared to conventional DVT prophylaxis approaches. In addition, it will add new values and benefits to public healthcare by eliminating additional treatment costs arising from DVT-related complications, increasing therapists' productivity (especially given growing manpower constraints and greying population), optimizing therapy time, and ultimately saving precious lives.

Among those diagnosed with DVT, 10-30% dies within 1 month of diagnosis (Beckman et al., 2010), and worldwide 600,000-800,000 people die annually (worldthrombosisday.org). This research seeks to lower DVT risk through a safe non-drug-based approach by continuously moving the ankle joint into dorsiflexion-plantarflexion using soft robotics. Current alternatives to prevent DVT include pharmacological prophylaxis such as anticoagulant drugs, mechanical prophylaxis such as intermittent pneumatic compression devices and compression stockings, and the basic therapist-assisted exercises to prevent ankle joint contractures. Pharmacological prophylaxis can improve venous blood flow and prevent DVT, but run the risk of detrimental side effects like excessive bleeding. Mechanical prophylaxis can provide passive or automated stimulation to the calf tissue, but have been reported to deliver limited efficacy in improving venous blood flow and preventing DVT. Considering the data from the United States and United Kingdom, the annual spending incurred due to direct and indirect costs resulting from DVT is approximated to be US$2-10 billion and this ranges from US$7,594-US$16,644 per patient (Spyropoulos and Lin, 2007). Therefore, by implementing the robotic sock device, the investigators hope to enable clinicians to focus on treating patients towards stroke recovery without worrying about other complications.

Joint contractures, usually defined as limited passive range of joint motion are common in people with neurological conditions such as stroke or spinal cord injury. The risk factors for joint contractures are not well understood; however, immobility seems to be the most important factors. Joint contractures, especially in the ankle joints, may impede the ability to walk and cause loss of balance, high risk of falls and restricted participation in social activities. The frequency of ankle contractures in hospitalized patients varies with prevalence rates ranging from 24 % to 44 %.

ELIGIBILITY:
Inclusion Criteria:

- Ischemic or haemorrhagic stroke patients with severe lower limb weakness (MRC scale <3) in flexors and extensors of knee and ankle

Exclusion Criteria:

* Medically unstable patients
* Queried pulmonary embolism (PE) / deep vein thrombosis (DVT) cases
* Limited range of motion in ankle and foot including equinus or club foot deformity
* Lower limb dermatitis, ulcer or open wound
* Severe spasticity of ankle (modified Ashworth scale >2)
* Pregnancy

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Presence of DVT | 4 weeks
  The primary outcome is a presence of DVT detected on a screening compression duplex ultrasonography
Ankle range of motion | 4 weeks
  Measurement of the range of motion of the ankle joint to determine the effect on joint contracture

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Beckman MG, Hooper WC, Critchley SE, Ortel TL. Venous thromboembolism: a public health concern. Am J Prev Med. 2010 Apr;38(4 Suppl):S495-501. doi: 10.1016/j.amepre.2009.12.017. PMID 20331949
- [Background] Roderick P, Ferris G, Wilson K, Halls H, Jackson D, Collins R, Baigent C. Towards evidence-based guidelines for the prevention of venous thromboembolism: systematic reviews of mechanical methods, oral anticoagulation, dextran and regional anaesthesia as thromboprophylaxis. Health Technol Assess. 2005 Dec;9(49):iii-iv, ix-x, 1-78. doi: 10.3310/hta9490. PMID 16336844
- [Background] Mazzone C, Chiodo GF, Sandercock P, Miccio M, Salvi R. Physical methods for preventing deep vein thrombosis in stroke. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD001922. doi: 10.1002/14651858.CD001922.pub2. PMID 15495020
- [Background] Spyropoulos AC, Lin J. Direct medical costs of venous thromboembolism and subsequent hospital readmission rates: an administrative claims analysis from 30 managed care organizations. J Manag Care Pharm. 2007 Jul-Aug;13(6):475-86. doi: 10.18553/jmcp.2007.13.6.475. PMID 17672809